CLINICAL TRIAL: NCT03331757
Title: Determination of the Glycemic Index and Glycemic Load of Six Greek Honey Grades
Brief Title: Determination of Glycemic Index of Six Greek Honey Grades
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agricultural University of Athens (Other)
Responsible Party: Principal Investigator, Aimilia Papakonstantinou, Primary investigator, Agricultural University of Athens
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 1254
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Potential Abnormality of Glucose Tolerance; Appetitive Behavior
MeSH Terms: conditions — Appetitive Behavior | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: Eleven healthy participants consumed in random order 50g available carbohydrates as glucose (tested three times) and 50g available carbohydrates as fir, chestnut, healther, thyme, pine, citrus, tested once, on separate occasions
Who Masked: Participant, Investigator
Masking Description: Participants were assigned to the interventions using a sequence of random numbers extracted from computer software. A researcher not involved with the collection and the analysis of the scientific data, was responsible for the randomization of the volunteers to the intervention days examining the test foods. All test meals (glucose and honeys) were diluted in 300ml water and were served in dark paper cups covered with a lid in order to achieve double blind conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Glucose as reference food (Experimental): Eleven metabolically healthy, normal weight subjects (male: 2, female: 9) after 10-14 hr fast, consumed 50g available carbohydrate from D-glucose, tested three times, in different weeks as reference food along with 300ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min. The first glucose sample was taken exactly 15min after the first drink.
  Interventions: Other: Glucose as reference food; Other: Fir honey; Other: Heather honey; Other: Citrus honey; Other: Pine honey; Other: Thyme honey; Other: Chestnut honey
- Fir honey (Experimental): Eleven metabolically healthy, normal weight subjects (male: 2, female: 9) after 10-14 hr fast, consumed 50g available carbohydrate from fir honey, tested once, along with 300ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min. The first glucose sample was taken exactly 15min after the first drink.
  Interventions: Other: Glucose as reference food; Other: Fir honey; Other: Heather honey; Other: Citrus honey; Other: Pine honey; Other: Thyme honey; Other: Chestnut honey
- Heather honey (Experimental): Eleven metabolically healthy, normal weight subjects (male: 2, female: 9) after 10-14 hr fast, consumed 50g available carbohydrate from heather honey, tested once, along with 300ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min. The first glucose sample was taken exactly 15min after the first drink.
  Interventions: Other: Glucose as reference food; Other: Fir honey; Other: Heather honey; Other: Citrus honey; Other: Pine honey; Other: Thyme honey; Other: Chestnut honey
- Citrus honey (Experimental): Eleven metabolically healthy, normal weight subjects (male: 2, female: 9) after 10-14 hr fast, consumed 50g available carbohydrate from citrus honey, tested once, along with 300ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min. The first glucose sample was taken exactly 15min after the first drink.
  Interventions: Other: Glucose as reference food; Other: Fir honey; Other: Heather honey; Other: Citrus honey; Other: Pine honey; Other: Thyme honey; Other: Chestnut honey
- Pine honey (Experimental): Eleven metabolically healthy, normal weight subjects (male: 2, female: 9) after 10-14 hr fast, consumed 50g available carbohydrate from pine honey, tested once, along with 300ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min. The first glucose sample was taken exactly 15min after the first drink.
  Interventions: Other: Glucose as reference food; Other: Fir honey; Other: Heather honey; Other: Citrus honey; Other: Pine honey; Other: Thyme honey; Other: Chestnut honey
- Thyme honey (Experimental): Eleven metabolically healthy, normal weight subjects (male: 2, female: 9) after 10-14 hr fast, consumed 50g available carbohydrate from thyme honey, tested once, along with 300ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min. The first glucose sample was taken exactly 15min after the first drink.
  Interventions: Other: Glucose as reference food; Other: Fir honey; Other: Heather honey; Other: Citrus honey; Other: Pine honey; Other: Thyme honey; Other: Chestnut honey
- Chestnut honey (Experimental): Eleven metabolically healthy, normal weight subjects (male: 2, female: 9) after 10-14 hr fast, consumed 50g available carbohydrate from chestnut honey, tested once, along with 300ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min. The first glucose sample was taken exactly 15min after the first drink.
  Interventions: Other: Glucose as reference food; Other: Fir honey; Other: Heather honey; Other: Citrus honey; Other: Pine honey; Other: Thyme honey; Other: Chestnut honey

INTERVENTIONS:
Other: Glucose as reference food — Eleven subjects (male: 2, female: 9) consumed 50g glucose diluted in 300ml water, tested three times, in different weeks, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min.
Other: Fir honey — Eleven subjects (male: 2, female: 9) consumed 50g available carbohydrates of fir honey diluted in 300ml water, tested once, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min.
Other: Heather honey — Eleven subjects (male: 2, female: 9) consumed 50g available carbohydrates of heather honey diluted in 300ml water, tested once, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min.
Other: Citrus honey — Eleven subjects (male: 2, female: 9) consumed 50g available carbohydrates of citrus honey diluted in 300ml water, tested once, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min.
Other: Pine honey — Eleven subjects (male: 2, female: 9) consumed 50g available carbohydrates of pine honey diluted in 300ml water, tested once, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min.
Other: Thyme honey — Eleven subjects (male: 2, female: 9) consumed 50g available carbohydrates of thyme honey diluted in 300ml water, tested once, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min.
Other: Chestnut honey — Eleven subjects (male: 2, female: 9) consumed 50g available carbohydrates of chestnut honey diluted in 300ml water, tested once, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min.

SUMMARY:
This study determined the glycemic index and glycemic load of six Greek honey varieties

DETAILED DESCRIPTION:
This randomized, double-blind, cross-over study investigated the glycemic response to six Greek honey grades differing in floral source and carbohydrate composition. Isoglucidic test meals (50g available carbohydrate) and 50g glucose reference were given to 11 clinically and metabolically healthy, fasting individuals (27±7 years; 9 women; BMI 24±4kg/m2), in random order. GI was calculated using the FAO/WHO method. Capillary blood glucose samples were collected at 0,15,30,45,60,90-and-120min. Salivary insulin samples were collected at 0,60-and-120min. Subjective appetite ratings (hunger, fullness and desire to eat) were assessed by visual analogue scales (VAS, 100mm) at baseline and 120min.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* non-smoking
* individuals with normal body mass index (between 18.5 and 24.9 kg/m2)

Exclusion Criteria:

* coronary heart disease
* diabetes mellitus
* kidney disease
* liver conditions
* endocrine conditions
* gastrointestinal disorders
* pregnancy
* lactation,
* competitive sports
* alcohol
* drug dependency

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2017-02-12 (Actual); Primary Completion 2017-04-12 (Actual); Study Completion 2017-09-02 (Actual)

PRIMARY OUTCOMES:
Capillary blood glucose responses | 2 hours
  Clinically useful change in capillary blood glucose, defined as the restoration of glucose within normal limits during the 2hr glucose tolerance test.

SECONDARY OUTCOMES:
Subjective appetite rating | 2 hours
  Useful change in subjective appetite using visual analogue scales (VAS, 100 mm, given in the form of booklet, one scale per page) before and 2hr after consumption of six Greek honey grades.

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Papakonstantinou, PhD, Principal Investigator — Agricultural University of Athens
Locations (1):
- Agricultural University of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: No